CLINICAL TRIAL: NCT04220658
Title: The NAD+ Baseline Study: a Biomarker-based Study to Evaluate Correlations Between Epigenetic Aging and NAD+ Levels in Healthy Volunteers
Brief Title: Biomarker Study to Evaluate Correlations Between Epigenetic Aging and NAD+ Levels in Healthy Volunteers
Status: Suspended | Type: Observational
Why Stopped: COVID-19
Sponsor: Elysium Health (Industry)
Collaborators: Duke Clinical Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Baseline Study
Record Dates: First submitted 2020-01-03; First posted 2020-01-07 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Epigenetics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples retained for 3 months, with potential for extraction of DNA from whole blood and/or saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biomarker study — Biomarkers of aging including NAD+ levels in whole blood, interleukins, inflammatory cytokines, growth factors, omega-3 polyunsaturated fatty acids, and patterns in DNA methylation

SUMMARY:
This is a single center, prospective study to evaluate correlations between epigenetic aging (as measured via DNA methylation) and NAD+ levels in healthy volunteers.

DETAILED DESCRIPTION:
This biomarker study consists of a single outpatient visit to the research unit. At this visit, eligibility will be assessed and biomarker samples (blood, saliva and urine) will be collected from subjects meeting eligibility criteria. Consenting subjects with clinically significant screening lab values may be excluded from the study after biomarker sample collection (i.e., clinical lab test results will become available after the biomarker sample collection). The prescribing of drugs to humans will not be part of this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females between 25 - 80 (inclusive) years of age
2. Able and willing to provide written consent, follow instructions to complete study questionnaire(s) and assessments
3. Peripheral venous access sufficient for blood draw

Exclusion Criteria:

1. History of any significant chronic disease including renal, liver, endocrine, inflammatory, cardiovascular, gastro-intestinal, neurological, psychiatric, neoplastic, or metabolic disease, unless well controlled (defined as stable medication regimen) for at least 90 days prior to screening. Clinical significance of active disease will be assessed by the Qualified Investigator to determine eligibility.
2. Clinically significant, unstable or untreated medical disorders including recent myocardial ischemia or infarction, unstable angina, uncontrolled hypertension, AIDS, malignancy, epilepsy, and recent cerebrovascular disease that required a change in management or hospitalization within the last 90 days.
3. Subjects with or who have recently experienced a traumatic injury, infections or undergone major surgery at the discretion of the Qualified Investigator
4. Donation or receipt of blood products within 90 days.
5. Clinically significant vital sign or physical examination abnormality at the discretion of the Qualified Investigator.
6. Subjects with history of pellagra or niacin deficiency
7. Alcohol use >2 standard alcoholic drinks per day within the past month
8. History of alcoholism or drug abuse within 1 year prior to screening
9. Use of medical marijuana or products containing cannabinoids in the 14 days prior to screening.
10. Use of lipid lowering agents (including fish oil) unless the dose has been stable for greater than 90 days prior to screening.
11. Use of natural health products containing nicotinamide riboside or niacin exceeding the RDA (16mg/day for males and 14mg/day for females) within 14 days prior to Screening. Potential participants will be asked to bring all supplements for evaluation at time of screening.
12. History of or current diagnosis of any cancer (except for successfully treated basal or squamous cell carcinoma of the skin) diagnosed less than 5 years prior to screening. Volunteers with cancer in full remission and more than 5 years after diagnosis are acceptable.
13. Has participated in any clinical trial with an investigational medicinal product within the past two months prior to the first dose in the current study
14. Clinically significant abnormal laboratory results at screening
15. Any other condition which in the Investigator's opinion may adversely affect the participant's ability to complete the study or its measures or which may pose significant risk to the participant
16. Consumption of non-water beverage or food within approximately 8 hours of sample collection

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals between 25-80 years of age
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2019-12-19 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-03 (Estimated)

PRIMARY OUTCOMES:
Correlation between biological age, calculated using DNA isolated from blood, and circulating NAD+ levels | At baseline

SECONDARY OUTCOMES:
Correlations between biological age, calculated using DNA isolated from saliva, and circulating NAD+ levels | At baseline
Correlations between biological age, calculated using DNA isolated from blood and saliva, and Omega-3 levels in blood | At baseline

OTHER OUTCOMES:
Age related markers in blood and urine | At baseline
  Correlations between biological age, calculated from DNA isolated from blood and saliva, and the following age-related markers observed in blood and urine:
  * Cellular senescence, proliferation and inflammation: CD3+ and p16INK4a+ T lymphocytes, TNF-α R1, IL-6, IL-8, IL-10, C-reactive protein, eotaxin, activin A, myostatin.
  * NAD-related biomarkers: CD38
  * Cellular health and bioenergetics: mitochondrial DNA and nuclear DNA

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Guptill, MD, Principal Investigator — Duke Early Phase Clinical Research/DCRI
Locations (1):
- Duke Early Phase Clinical Research, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No